CLINICAL TRIAL: NCT04137276
Title: Effect of Intravenous Vitamin C on Sequential Organ Failure Assessment (SOFA) Score Among Septic Patients: Randomized Controlled Trial
Brief Title: Effect of Intravenous Vitamin C on SOFA Score Among Septic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, Staff Lecturer at Department of Anesthesiology and Intensive Care, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes 39
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Sepsis
Keywords: sepsis; intravenous vitamin C; SOFA score
MeSH Terms: conditions — Sepsis | interventions — Ascorbic Acid; Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin C and thiamine (Experimental): patients who received intravenous vitamin C and thiamine
  Interventions: Drug: vitamin C, vitamin B1
- thiamine (Active Comparator): patients who received thiamine
  Interventions: Drug: vitamin B1

INTERVENTIONS:
Drug: vitamin C, vitamin B1 — vitamin C 1,5 g/6 hours IV + thiamine 200 mg/12 hours for 3 days
  Other Names: group A
  Arms: vitamin C and thiamine
Drug: vitamin B1 — thiamine 200 mg/12 hours for 3 days
  Other Names: group B
  Arms: thiamine

SUMMARY:
This study aimed to explore the effect of intravenous (IV) vitamin C on sequential organ failure assessment (SOFA) score among septic patients in intensive care unit (ICU).

DETAILED DESCRIPTION:
"This study was approved by the Ethics and Research Committee of Universitas Indonesia. This study was a randomized clinical trial held from April to July 2019 in Cipto Mangunkusumo Hospital. 33 patients that met the inclusion criteria were included in the study. Subjects were divided into two groups: group A (intervention group, n = 18) received parenteral infusions of 1,5 g/6 hours of vitamin C and 200 mg thiamine, while group B (control group, n = 15) received 200 mg thiamine only. baseline demographic data was recorded on the first day. SOFA score was recorded at baseline, 24 hours, 48 hours, and 72 hours after treatment. Data were analyzed using SPSS (Statistical Package for Social Sciences) software."

ELIGIBILITY:
Inclusion Criteria:

* patients with sepsis diagnosis based on sepsis-3 criteria in the ICU in between 6 hours to 24 hours post resuscitation after sepsis diagnosis

Exclusion Criteria:

* patients with chronic kidney problems on haemodialysis,
* patients with kidney stones or kidney problem within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | 3 months
  Sequential Organ Failure Assessment (SOFA) score score measured at several specified times. higher score indicates higher mortality in septic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Adhrie Sugiarto, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Carr AC, Shaw GM, Fowler AA, Natarajan R. Ascorbate-dependent vasopressor synthesis: a rationale for vitamin C administration in severe sepsis and septic shock? Crit Care. 2015 Nov 27;19:418. doi: 10.1186/s13054-015-1131-2. PMID 26612352
- [Result] Bagshaw SM, George C, Bellomo R; ANZICS Database Management Committee. Early acute kidney injury and sepsis: a multicentre evaluation. Crit Care. 2008;12(2):R47. doi: 10.1186/cc6863. Epub 2008 Apr 10. PMID 18402655
- [Result] Bellomo R, Kellum JA, Ronco C, Wald R, Martensson J, Maiden M, Bagshaw SM, Glassford NJ, Lankadeva Y, Vaara ST, Schneider A. Acute kidney injury in sepsis. Intensive Care Med. 2017 Jun;43(6):816-828. doi: 10.1007/s00134-017-4755-7. Epub 2017 Mar 31. PMID 28364303
- [Result] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003
- [Result] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Result] Oudemans-van Straaten HM, Elbers PWG, Spoelstra-de Man AME. How to Give Vitamin C a Cautious but Fair Chance in Severe Sepsis. Chest. 2017 Jun;151(6):1199-1200. doi: 10.1016/j.chest.2017.01.008. Epub 2017 Apr 7. No abstract available. PMID 28599924
- [Result] Moskowitz A, Andersen LW, Cocchi MN, Karlsson M, Patel PV, Donnino MW. Thiamine as a Renal Protective Agent in Septic Shock. A Secondary Analysis of a Randomized, Double-Blind, Placebo-controlled Trial. Ann Am Thorac Soc. 2017 May;14(5):737-741. doi: 10.1513/AnnalsATS.201608-656BC. PMID 28207287
- [Result] Abiles J, de la Cruz AP, Castano J, Rodriguez-Elvira M, Aguayo E, Moreno-Torres R, Llopis J, Aranda P, Arguelles S, Ayala A, de la Quintana AM, Planells EM. Oxidative stress is increased in critically ill patients according to antioxidant vitamins intake, independent of severity: a cohort study. Crit Care. 2006;10(5):R146. doi: 10.1186/cc5068. PMID 17040563
- [Result] Galley HF, Howdle PD, Walker BE, Webster NR. The effects of intravenous antioxidants in patients with septic shock. Free Radic Biol Med. 1997;23(5):768-74. doi: 10.1016/s0891-5849(97)00059-2. PMID 9296454